CLINICAL TRIAL: NCT00004404
Title: Study of Clotrimazole and Hydroxyurea in Patients With Sickle Cell Syndromes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: 199/13288; CH-B-97-052; CH-B-FDR001022
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1998-05

CONDITIONS: Sickle Cell Anemia
Keywords: genetic diseases and dysmorphic syndromes; hematologic disorders; rare disease; sickle cell anemia
MeSH Terms: conditions — Anemia, Sickle Cell; Genetic Diseases, Inborn; Hematologic Diseases; Rare Diseases | interventions — Clotrimazole; Hydroxyurea

INTERVENTIONS:
Drug: clotrimazole
Drug: hydroxyurea

SUMMARY:
OBJECTIVES:

Determine the effectiveness of the combined use of clotrimazole and hydroxyurea on a specific panel of red cell characteristics in patients with sickle cell syndromes.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients receive oral hydroxyurea either once or twice daily plus oral clotrimazole twice daily after meals for 6 months. Patients are assessed at 3 and 6 months during treatment.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Sickle cell syndromes characterized by vaso-occlusive crises sufficiently severe to require prophylactic therapy Three or more crises per year sufficiently severe to require hospitalization Stable dose of hydroxyurea for at least 4 months required --Prior/Concurrent Therapy-- No treatment with any other antisickling agents within the past 4 months Biologic therapy: No transfusion within 90 days No concurrent chronic transfusions allowed (defined as more than one transfusion per month for 2 or more months) Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: No chronic medications that alter neurologic, renal, or hepatic functions

* Patient Characteristics-- Performance status: Karnofsky 70-100% Hematopoietic: WBC within normal limits Platelet count within normal limits Hepatic: No history of chronic liver disease Bilirubin less than 2 times normal SGOT and SGPT less than 2.5 times normal No severe hepatic damage Renal: Creatinine within normal limits No severe renal damage Neurologic: No severe neurologic impairment No recent or progressive neurologic impairment Other: Not pregnant Fertile patients must use effective contraception No allergies to hydroxyurea or clotrimazole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 1997-04; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Brugnara, Study Chair — Boston Children's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Children's Hospital - Boston, Boston, Massachusetts